CLINICAL TRIAL: NCT05095896
Title: The Serum Lipid Profiles in Immune Thrombocytopenia: a Retrospective Study
Brief Title: The Serum Lipid Profiles in ITP: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Ming Hou (Other)
Responsible Party: Sponsor-Investigator, Ming Hou, Manager, Shandong University
Organization: Shandong University (Other)
Other Study IDs: lipid in ITP
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ITP patients — ITP patients were enrolled in this study based on Chinese consensus of ITP.12 Patients were excluded as (1) receiving platelet transfusion within 7 days or ITP-related medication within 3 months (2) treated with lipid-lowing agents, including statins, fibrates, niacin, bile sequestrant resins, ezetimibe and so on.

SUMMARY:
The project was retrospectively undertaking by Qilu Hospital of Shandong University in China. In order to investigate the correlations between platelet indices, serum lipids and bleeding symptoms in ITP.

DETAILED DESCRIPTION:
Background: Immune thrombocytopenia (ITP) is an autoimmune hemorrhagic disease characterized by increased platelet destruction and impaired thrombopoiesis. Platelet indices changes depending on the morphology and volume of platelets. Serum lipids have been found to affect platelet formation and activity in certain diseases, thus induce the corresponding variation of platelet indices.

Objectives: To investigate the correlations between platelet indices, serum lipids and bleeding symptoms in ITP.

Methods: The clinical data from 457 ITP patients were retrospectively collected and analyzed, including platelet indices, serum lipids, hemorrhage and therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for immune thrombocytopenia.

Exclusion Criteria:

* (1) receiving platelet transfusion within 7 days or ITP-related medication within 3 months (2) treated with lipid-lowing agents, including statins, fibrates, niacin, bile sequestrant resins, ezetimibe and so on.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 457 ITP patients at Department of Hematology of Qilu Hospital were enrolled in this study based on Chinese consensus of ITP.12 Patients were excluded as (1) receiving platelet transfusion within 7 days or ITP-related medication within 3 months (2) treated with lipid-lowing agents, including statins, fibrates, niacin, bile sequestrant resins, ezetimibe and so on.
Sampling Method: Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Platelet count at 1 month after initial therapy | 1 month
  Platelet count was tested at 1 month after initial therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu P, Han S, Hou M, Zhao Y, Xu M. The serum lipid profiles in immune thrombocytopenia: Mendelian randomization analysis and a retrospective study. Thromb J. 2023 Oct 13;21(1):107. doi: 10.1186/s12959-023-00551-x. PMID 37833799